CLINICAL TRIAL: NCT02786862
Title: 1:1 Proportion Ventilation With a Unique Device for Independent Lung Ventilation Using a Double-Lumen Tube in the Supine and Lateral Decubitus Positions. A Pilot Study
Brief Title: A Unique Device for Independent Lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lublin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MULublin
Record Dates: First submitted 2016-04-11; First posted 2016-06-01 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Anesthesia
Keywords: mechanical ventilation; independent ventilation; ventilation/perfusion mismatch; thoracic anesthesia
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ventilation (Experimental): Measurements were made for conventional and independent at 1:1 proportion ventilation in supine position; then independent ventilation was discontinued and patient was moved to right or left decubitus position due to left or right lung surgery. Then were made measurements for conventional anaesthetic practices and followed independent at 1:1, 2:1, 3:1, 5:1 proportions ventilation routines. Constantly were monitored expired volume, peak respiratory pressure, dynamic compliance separately for each lung. Measurements covered also hemodynamic (MAP, HR) and oxygenation (SpO2). These attributes were documented at each point of the study. Subsequently, the control system was disconnected and performed typical anaesthetic procedures for thoracic surgery with a one-lung ventilation procedure.
  Interventions: Other: independent ventilation

INTERVENTIONS:
Other: independent ventilation — comparison conventional and independent 1:1 ventilation

SUMMARY:
Adequate blood oxygenation and ventilation/perfusion matching should be the main goal of anaesthetic and intensive care management. At present, the sole method of improving gas exchange restricted by ventilation/perfusion mismatching is independent ventilation with two ventilators. Recently, however, a unique device has been developed, enabling ventilation of independent lungs in 1:1, 2:1, 3:1, and 5:1 proportions. The main goal of the study was to evaluate the device's utility, precision and impact on biomechanical lung parameters during thoracic surgery under general anaesthesia with double lumen tube intubation. Secondly- to measure the gas distribution in supine and lateral decubitus position.

DETAILED DESCRIPTION:
Anaesthetic management:

One hour before thoracic surgery, the patient-subjects received diazepam 0.15 mg kg-1 as premedication. After arriving at the operating theatre, standard monitoring system practices was applied, including heart rate (HR), systolic arterial pressure (SAP), diastolic arterial pressure (DAP), mean arterial pressure (MAP), and pulse oximetry (SpO2). Moreover, an intra-vein cannula was placed, and the infusion of multi-electrolytic fluid 5-10 ml kg-1 h-1 was started. After pre-oxygenation, atropine 0.5 mg and fentanyl 3 µg kg-1 were given, and the induction of anaesthesia with thiopentone 5-7 mg kg-1 was started. Suxamethonium was administered for neuromuscular blockade, and bronchial intubation with a Robertshow double lumen tube was performed. The left bronchus was intubated for right lung surgery, and the right bronchus was intubated for left lung surgery. Tube placement was checked via auscultation and fiberscope. Anaesthesia was maintained with sevoflurane, additional fentanyl doses were used if needed, and neuromuscular blockade was obtained with vecuronium 0.1 mg kg-1. Additionally, 0.1 mg kg-1 dose of morphine was given subcutaneously for postoperative pain control. Patients were also ventilated with O2 (oxygen) and AIR (air) mixture, using the following settings: volume control intermittent positive pressure ventilation, FiO2 (oxygen fraction) 0.4, Vt (tidal volume) 6-10 ml/kg, and f (frequency) 12-15 /min. Furthermore, end tidal CO2 (carbon dioxide) was monitored due to normocapnia maintenance (4.0-5.3 kPa). At the end of surgery, intercostal blockade was brought about with 0.5% bupivacaine, with 5 ml for each nerve. Finally, the neuromuscular blockade was reversed with neostigmine 0.04 mg kg-1 and with atropine 0.01 mg kg-1.

After anaesthesia stabilisation, the unique control system was used, called the 'tidal volume divider'. This device was placed between the anaesthetic machine and the double lumen tube of the patient. This control system enables conventional ventilation (without any intervention from the control system, as the settings are defined on the ventilator), as well as independent ventilation with division of the tidal volume between the lungs in proportions of 1:1, 2:1, 3:1, and 5:1. It also enables PEEP (selective positive end-expiratory pressure) application to each lung. With independent ventilation, settings such as frequency, tidal volume and inspiration time are defined by ventilator, and this system only controls the direction of tidal volume to each lung (as the control system is a flow divider) by using a differential pneumatic resistor. It also enables dependent and non-dependent lung ventilation in the lateral decubitus positions. Furthermore, the system monitors the expired volume, airway pressure and dynamic compliance of each lung. This device was described and tested on mechanical lung models with a variety of lung model mechanics (compliance, resistance) and ventilation parameters (frequency, tidal volume). It was also tested clinically for its safety during our previous study. The system was invented, developed and patented by a group of Polish engineers from the Nałęcz Institute of Biocybernetics and Biomedical Engineering, the Polish Academy of Sciences, Poland.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II patients who underwent elective thoracic surgery under general anaesthesia, with double lumen tube intubation and one lung ventilation during surgical procedure.

Exclusion Criteria:

* All patients with asthma or chronic obstructive pulmonary disease, history of thoracotomy, assessed as ASA III, with difficult airway conditions, kyphoscoliosis or other alterations of chest wall or severe obesity were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Tidal volume distribution during conventional and independent in 1:1 proportion ventilation in supine, left and right decubitus positions. | up to 12 months
  tidal volume

SECONDARY OUTCOMES:
Peak respiratory pressure measuring during conventional and independent in 1:1 proportion ventilation in supine, left and right decubitus positions. | up to 12 months
  peak respiratory pressure
Dynamic compliance measuring during conventional and independent in 1:1 proportion ventilation in supine, left and right decubitus positions. | up to 12 months
  dynamic compliance

OTHER OUTCOMES:
Impact of supine to left and supine to right decubitus position changes on tidal volume distribution during conventional and independent in 1:1 proportion ventilation. | up to 12 months
  tidal volume
Impact of supine to left and supine to right decubitus position changes on peak respiratory pressure, during conventional and independent in 1:1 proportion ventilation. | up to 12 months
  peak respiratory pressure
Impact of supine to left and supine to right decubitus position changes on dynamic compliance during conventional and independent in 1:1 proportion ventilation. | up to 12 months
  dynamic compliance

CONTACTS AND LOCATIONS:
Overall Officials: Slawomir Sawulski, M.D., Ph.D., Principal Investigator — Medical University of Lublin, Poland

IPD SHARING:
Plan to Share IPD: Yes
Row data will be attached as supplementary files during publication process
Supporting Information: Study Protocol
Time Frame: Row data will be attached as supplementary files during publication process
Access Criteria: Data will be available for everybody

REFERENCES:
- [Background] Darowski M, Englisz M. Artificial ventilation of the lungs for emergencies. Front Med Biol Eng. 2000;10(3):177-83. doi: 10.1163/15685570052062576. PMID 11014679
- [Background] Sawulski S, Nestorowicz A, Sawicki M, Kowalczyk M, Ston M. [Independent lung ventilation during general anaesthesia--preliminary report]. Anestezjol Intens Ter. 2010 Jan-Mar;42(1):6-10. Polish. PMID 20608207